CLINICAL TRIAL: NCT00612547
Title: Assessment of the Use of Fixed Doses of Artesunate Plus Amodiaquine Combination for the Home Management of Presumed Malaria in Malagasy Children
Brief Title: ACT for the Home Management in Malagasy Children
Status: Completed | Type: Observational
Sponsor: National Malaria Control Programme, Madagascar (Other Government)
Collaborators: Population Services International (Other); Reggio Terzo Mondo (Unknown); Santé Net (Unknown); Inter Aide Santé, (Unknown); Adventist Development and Relief Agency (Other); SAF FJKM (Unknown); Sanofi (Industry); Institut Pasteur de Madagascar (Other)
Responsible Party: Didier Ménard, Head of the Malaria Research Unit, Institut Pasteur de Madagascar
Other Study IDs: ACTComMada
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Fever; Suspected Malaria
Keywords: Protozoan Infections; Communicable Diseases; Malaria Infection; Malaria, falciparum; Malaria, vivax; Artesunate Amodiaquine
MeSH Terms: conditions — Fever; Protozoan Infections; Communicable Diseases; Malaria, Falciparum; Malaria, Vivax | interventions — Artesunate; Amodiaquine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Children under the age of five years (2 months to 5 years) residing in the zone covered by the community-based service provider throughout the entire follow-up period
  Interventions: Drug: Artesunate + Amodiaquine Fixed Dose Combination (CoArsucam)

INTERVENTIONS:
Drug: Artesunate + Amodiaquine Fixed Dose Combination (CoArsucam) — Tablet:
  Children aged between 2 and 11 months: Artesunate 25 mg + Amodiaquine 67.5 mg et Children aged between 12 and 59 months: Artesunate 50 mg + Amodiaquine 135 mg Per os one intake per day/3 day

SUMMARY:
The purpose of this study is to assess the feasibility, the acceptability and the effectiveness of the use of the Artesunate + Amodiaquine Fixed Dose Combination for the home management of presumed malaria in Malagasy children by the community-based service providers.

DETAILED DESCRIPTION:
Primary objective

To assess the feasibility, the acceptability and the effectiveness of the use of the Artesunate + Amodiaquine Fixed Dose Combination for the home management of presumed malaria in Malagasy children by the community-based service providers

Secondary objectives

To assess the reliability of the use of the malaria rapid diagnostic tests (RDT) by the community-based service providers in the Malagasy home management strategy

To assess the frequency of short-term and long-term side effects of the Artesunate + Amodiaquine Fixed Dose Combination used for the home management of presumed malaria in Malagasy children by the community-based service providers

To assess the real burden of the malaria in children under the age of five years in 2 different epidemiological strata of Madagascar (central highlands and equatorial strata)

Type of study

Follow-up of a cohort of 1200 children under the age of five years during 1 year

Studied population

All children under the age of five years (2 months to 5 years) having fever and consulting the community-based service provider, residing in the zone covered by the community-based service provider throughout the entire follow-up period Investigators Four community-based service providers, four field physicians and two supervisors number of district: 2 (Moramanga and Manakara)

condition: fever intervention: artesunate + amodiaquine phase: phase IV

ELIGIBILITY:
Inclusion Criteria:

* All children under the age of five years (2 months to 5 years) having fever and consulting the community-based service provider, residing in the zone covered by the community-based service provider throughout the entire follow-up period, having signed an informed consent

Exclusion Criteria:

* Children with no informed consent

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Assessment of the councils delivered by the community-based service provider to the parents or guardians of children and assessment of the observance of the treatment given by the parents or guardians. | one year

SECONDARY OUTCOMES:
To assess the Artesunate + Amodiaquine Fixed Dose Combination in term of effectiveness, tolerance, safety:; the reliability of the RDT; the real burden of the malaria in children under the age of five years in 2 different epidemiological strata. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Ramarosandratana, MD, Study Chair — National Malaria Control Programme
Locations (1):
- Institut Pasteur, Paris, France

REFERENCES:
- [Derived] Ratsimbasoa A, Ravony H, Vonimpaisomihanta JA, Raherinjafy R, Jahevitra M, Rapelanoro R, Rakotomanga Jde D, Malvy D, Millet P, Menard D. Management of uncomplicated malaria in febrile under five-year-old children by community health workers in Madagascar: reliability of malaria rapid diagnostic tests. Malar J. 2012 Mar 25;11:85. doi: 10.1186/1475-2875-11-85. PMID 22443344